CLINICAL TRIAL: NCT04566939
Title: A Long Term Follow-Up of Rotator Cuff Tear Patients Treated With Integrated Complementary and Alternative Medicine: Retrospective Chart Review and Survey Study
Brief Title: A Long Term Follow-Up of Rotator Cuff Tear Patients Treated With Integrated Complementary and Alternative Medicine
Status: Completed | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Other Study IDs: JS-CT-2020-11
Record Dates: First submitted 2020-09-24; First posted 2020-09-28 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator cuff tear, Korean medical treatment
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Phytotherapy; Acupuncture Therapy; Electroacupuncture; Cupping Therapy; Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Herbal medicine — Herbal medicine will be administered in water-based decoction (120ml) and dried powder (2g) form (Ostericum koreanum,Eucommia ulmoides, canthopanax sessiliflorus, Achyranthes japonica, Psoralea corylifolia, aposhnikovia divaricata, Cibotium barometz, Lycium chinense, Boschniakia rossica, Cuscuta chinensis, Glycinemax, Atractylodes japonica) at the physician's discretion.
  Other Names: Traditional herbal medicine
Procedure: Chuna manual medicine — Chuna is a Korean manual therapy directed at the spine and joints that incorporates various spinal manual medicine techniques for joint mobilization involving high-velocity, low amplitude thrusts to joints slightly beyond the passive range of motion and gentle force to joints within the passive range of movement. Chuna manual medicine will be administered to the shoulder at the physician's discretion.
  Other Names: Chuna manipulation
Procedure: Pharmacopuncture — Pharmacopuncture consisting of select herbal ingredients will be administered at Gyunwoo (LI15), Gyunryo(TE14), Ah-shi points and local acupuncture points using disposable injection needles (CPL, 1 cc, 26G x 1.5 syringe, Shinchang medical co., Korea) at the physician's discretion.
Procedure: Acupuncture — Acupuncture treatment will be administered using mainly proximal acupuncture points and Ah-shi points.
Procedure: Electroacupuncture — Electroacupuncture treatment will be administered using mainly proximal acupuncture points and Ah-shi points.
Procedure: Cupping — Cupping treatment will be administered at 1-2 points using mainly proximal acupuncture points and Ah-shi points.
Procedure: Herbal hot pack — Herbal hot pack treatment will be administered using mainly proximal acupuncture points and Ah-shi points.
Procedure: Physical therapy — The participants in the control group will be receive one or more physical therapy according to the physician's decision.
Procedure: Other intervention(s) — Patients will be allowed any other additional intervention(s) as deemed necessary regardless of type or dose, and patterns of use will be investigated and recorded as a pragmatic clinical study.

SUMMARY:
This study is a prospective observational trial. Data of 4 hospitals will be used to find out the efficacy of conservative treatment in rotator cuff tear.

DETAILED DESCRIPTION:
"Rotator cuff tear is known as its symptoms which are pain, limited shoulder range of motion(ROM), and the clicking sound of the shoulder.

On recent research by Health Insurance Review & Assessment Service, the number of rotator cuff tear patients has increased from 508155 to 704838 during 2013-2017. And also the research reported that the difference of effect between surgical treatments and non-surgical treatments was unremarkable. So in most cases, non-surgical treatments are applied primarily on rotator cuff tear except for some serious cases.

Physical therapy and medication are well known for the currently known non-surgical and conservative treatments, but research reported on the treatment of rotator cuff tear by using Korean medicine treatment so far has its weak level. Therefore, it is expected that this study will demonstrate the efficacy of the treatment of rotator cuff tear in Korean medicine treatment and will further pave the way for non-surgical treatment of rotator cuff tear.

Therefore, The investigators conducted an observational trial to analyze the effectiveness of Korean medicine treatment in rotator cuff tear. Retrospective data will be extracted using electronic medical records and computerized data of hospitalized patients. Based on this, investigators will conduct research in the form of a prospective survey and analyze the causal relationship and factors using the two data.

The hospital's medical records will be used to analyze the patient's condition during the hospitalization period and to determine the situation after the end of treatment through a questionnaire. The questionnaire will be developed after consultation with experts from the musculoskeletal system and related societies, and will be used for the questionnaire."

ELIGIBILITY:
Inclusion Criteria:

* Patients who had been hospitalized with symptoms of shoulder pain at Haeundae Jaseng Korean Medicine Hospital, Jaseng Korean Medicine Hospital, Bucheon Jaseng Korean Medicine Hospital and Daejeon Jaseng Korean Medicine Hospital from Jan 2015 to Mar 2020.
* Patients diagnosed with 'Rotation Cuff Tear' finding of the EMR imaging (T2-weighted MRI scan of Shoulder
* Patients who had been hospitalized more than 3 days
* Patients who are within age from 19 to 70

Exclusion Criteria:

* Patients who are hospitalized by traffic accident
* Patients who are diagnosed other serious shoulder injury that can cause shoulder pain(tumor of shoulder, acute fracture and dislocation of shoulder)
* Patients who had treated shoulder pain at Haeundae Jaseng Korean Medicine Hospital, Jaseng Korean Medicine Hospital, Bucheon Jaseng Korean Medicine Hospital and Daejeon Jaseng Korean Medicine Hospital in recent 6 months.
* Patients who are considered impossible to attend survey by investigators.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who ended up the hospitalization and treatment in Haeundae Jaseng Korean Medicine Hospital, Jaseng Korean Medicine Hospital, Bucheon Jaseng Korean Medicine Hospital, Daejeon Jaseng Korean Medicine Hospital
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain intensity scale: Numeric Rating Scale (NRS) | Finish survey by March 2021
  The investigators will survey Shoulder Pain intensity scale: Numeric Rating Scale (NRS) before hospitalization and after discharging from 4 hospitals(Haeundae Jaseng Korean Medicine Hospital, Jaseng Korean Medicine Hospital, Bucheon Jaseng Korean Medicine Hospital, and Daejeon Jaseng Korean Medicine Hospital.
  The score ranges from 0 to 10. The higher scores mean a worse outcome, and the lower scores mean a better outcome.

SECONDARY OUTCOMES:
Functional scale: Shoulder Pain and Disability Index (SPADI) | Finish survey by March 2021
  The investigators will survey Functional scale: Shoulder Pain and Disability Index (SPADI) of hospitalization period and after discharging in 4 hospitals(Haeundae Jaseng Korean Medicine Hospital, Jaseng Korean Medicine Hospital, Bucheon Jaseng Korean Medicine Hospital, and Daejeon Jaseng Korean Medicine Hospital).
5-Level Quality of life: EuroQol 5-Dimension (EQ-5D-5L) | Finish survey by March 2021
  The investigators will survey 5-Level Quality of life: EuroQol 5-Dimension (EQ-5D-5L) of hospitalization period and after discharging in 4 hospitals(Haeundae Jaseng Korean Medicine Hospital, Jaseng Korean Medicine Hospital, Bucheon Jaseng Korean Medicine Hospital, and Daejeon Jaseng Korean Medicine Hospital).
Patient Global Impression of Change (PGIC) | Finish survey by March 2021
  The investigators will survey Patient Global Impression of Change (PGIC) of hospitalization period and after discharging in 4 hospitals(Haeundae Jaseng Korean Medicine Hospital, Jaseng Korean Medicine Hospital, Bucheon Jaseng Korean Medicine Hospital, and Daejeon Jaseng Korean Medicine Hospital).

CONTACTS AND LOCATIONS:
Overall Officials: HYUN WOO CHO, PhD, Principal Investigator — Haeundae Jaseng Hospital of Korean Medicine
Locations (1):
- Haeundae Jaseng Hospital of Korean Medicine, Busan, South Korea

REFERENCES:
- [Derived] Yoo DH, Choi JY, Lee SG, Choi KW, Park HB, Kim H, Cho H, Kim SD, Kim D, Lee YJ, Park KS, Ha IH. Long-Term Follow-Up of Inpatients with Rotator Cuff Tear Who Received Integrative Korean Medicine Treatment: A Retrospective Analysis and Questionnaire Survey. Explore (NY). 2024 Mar-Apr;20(2):212-221. doi: 10.1016/j.explore.2023.08.005. Epub 2023 Aug 25. PMID 37689574